CLINICAL TRIAL: NCT00628472
Title: Novel Technique for Botulinum Toxin Injection to Minimize Patient Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, David M. Ozog, Chair-Dermatology, Henry Ford Health System
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB 4300
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Pain
Keywords: botulinum toxin a; botox; Decreasing botox injection pain; injections
MeSH Terms: conditions — Pain | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: botulinum type a — 12 Units total were injected into 6 sites in the glabellar complex to determine if injecting through the follicle versus a traditional approach would decrease patient discomfort
  Other Names: Botox

SUMMARY:
This single blinded randomized pilot study was performed on 21 Caucasian females to determine if injections through follicular openings were less painful than traditional injections for cosmetic botulinum toxin type A injections.

DETAILED DESCRIPTION:
Objective: To investigate whether injection of botulinum toxin type A is less painful if performed through follicular openings versus traditional non-specific approach.

Design: Prospective, randomized, single-blinded study.

Setting: Academic dermatology department.

Patients: A volunteer sample of twenty female patients aged 25-55 who had no prior history of botulinum toxin injection.

Intervention: Each patient received six randomized injections of botulinum toxin type A (Botox® Allergan). Two injections into the procerus muscle and two into each corrugator muscle. Three of the injections were performed through follicular openings and three were performed traditionally.

Main Outcome Measure: Patient discomfort on a 1-10 scale and direct comparison between the two injection techniques.

ELIGIBILITY:
Inclusion Criteria:

* Female
* No prior history of botulinum toxin
* Age 25-55

Exclusion Criteria:

* Male
* Prior history of botulinum toxin
* Neuromuscular disorders
* Aminoglycoside therapy

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2007-01; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Decrease pain on injection for treatment intervention assessed on a 10 point scale | At time of intervention

CONTACTS AND LOCATIONS:
Overall Officials: David M Ozog, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States